CLINICAL TRIAL: NCT04028518
Title: A PhaseⅡ, Multicenter, Prospective Randomised, Open Blinded Endpoint Study to Evaluate Safety and Efficacy of Injection for Recombinant Human Tissue Plasminogen Kinase Derivative in Treatment of Acute Ischemic Stroke.
Brief Title: A PhaseⅡ of Injection for Recombinant Human Tissue Plasminogen Kinase Derivative in Treatment of Acute Ischemic Stroke.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Angde Biotech Pharmaceutical Co., Ltd. (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD-RTL-202
Record Dates: First submitted 2019-06-13; First posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-06

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Injections; Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The high-dose group (Experimental): Experimental: r-PA Dose: stick 18 mg;
  Mode of admin:
  The high-dose group (18 mg + 18 mg) was divided into two intravenous injections. the first intravenous bolus injection of 18mg,after 30mins, the second intravenous bolus injection of 18 mg, Push slowly for more than 2mins each time.Subjects were closely monitored during the medication and within 24 hours of administration.
  Interventions: Drug: r-PA
- The low-dose group (Experimental): Experimental: r-PA Dose: stick 18 mg;
  Mode of admin:
  The low-dose group (12 mg + 12 mg) was divided into two intravenous injections, the first intravenous bolus injection of 12 mg, after 30mins, the second intravenous bolus injection of 12 mg, Push slowly for more than 2mins each time.Subjects were closely monitored during the medication and within 24 hours of administration.
  Interventions: Drug: r-PA
- Active Comparator: Alteplase (Experimental): Active Comparator: Alteplase Drug: Alteplase for Injection Dose:50mg;20mg
  Mode of admin:
  0.9 mg/kg (maximum dose of 90 mg) intravenous, 10% of which was injected intravenously within the first 1min, and the rest continued intravenous infusion for 1 h. Subjects should be closely monitored during the treatment period and within 24 hours of medication.Subjects were monitored according to the "Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke in China 2018".
  Interventions: Drug: Alteplase for Injection

INTERVENTIONS:
Drug: r-PA — Drug: r-PA Dose: stick 18 mg;
  Mode of admin:
  The high-dose group (18 mg + 18 mg) was divided into two intravenous injections. the first intravenous bolus injection of 18mg,after 30mins, the second intravenous bolus injection of 18 mg, Push slowly for more than 2mins each time.
  Other Names: Recombinant Human Tissue Plasminogen Kinase Derivative for Injection
  Arms: The high-dose group
Drug: r-PA — Drug: r-PA Dose: stick 18 mg;
  Mode of admin:
  The low-dose group (12 mg + 12 mg) was divided into two intravenous injections, the first intravenous bolus injection of 12 mg, after 30mins, the second intravenous bolus injection of 12 mg, Push slowly for more than 2mins each time.
  Other Names: Recombinant Human Tissue Plasminogen Kinase Derivative for Injection
  Arms: The low-dose group
Drug: Alteplase for Injection — Drug: Alteplase for Injection Dose:50mg; 20mg
  Mode of admin:
  0.9 mg/kg (maximum dose of 90 mg) intravenous, 10% of which was injected intravenously within the first 1min, and the rest continued intravenous infusion for 1 h.
  Other Names: Recombinant Human Tissue Plasminogen Active for Injection
  Arms: Active Comparator: Alteplase

SUMMARY:
The primary purpose of this trial is to compare the efficacy of different doses of investigator product and comparator product in patients with acute ischemic stroke in 4.5 Hours after stroke onset, and provide a basis of drug administration for phase Ⅲ clinical trial.

The secondary purpose of this trial is to compare the safety of different dose of investigational product and comparator product in patients with acute ischemic stroke in 4.5 hours afterstroke onset .

DETAILED DESCRIPTION:
This study is a multicenter, prospective randomised, open blinded endpoint study.

Patients with acute ischemic stroke need to undergo CT or MRI to exclude intracranial hemorrhage and perform NIHSS score before enrollment. Subjects who have passed the screening criteria according to the inclusion and exclusion criteria will be randomly assigned to low-dose test drugs, high-dose test drugs or reference drugs for thrombolytic therapy at a ratio of 1:1:1. The random stratification factor is the thrombolysis time window ("≤3h" vs "3~4.5h").

The start of administration of the study drug is recorded as 0h, CT or MRI and NIHSS score, laboratory test, and electrocardiogram were performed at 24 hours; NIHSS score was performed at 72 hours; NIHSS score，laboratory test and electrocardiogram were performed on the14th day(the start of administration is recorded as Day 1 ,then the 14th day after administration should be recorded as Day 15 ); mRS score and Barthel index score were performed on the 30th day (Day 31); mRS score and Barthel index score were performed on the 90th day (Day 91).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute ischemic stroke according to the WHO (World Health Organization) stroke diagnostic criteria, and symptoms of stroke have existed for at least 30mins, and there is no significant improvement before treatment；
* The symptoms of acute ischemic stroke are expected to be less than 4.5 hours after the time of acute ischemic stroke which is defined as the last time the patient function well;
* NIHSS score at the time of treatment: from 4 points to 24 points (including 4 points and 24 points);
* From the signing of informed consent form to 3 months of the last dose should be the absence of a birth plan and willing to take effective contraceptive measures;
* Understand and follow the research process, voluntarily participate, and sign an informed consent form (informed consent is voluntarily signed by the person or legal representative).

Exclusion Criteria:

* Weight >120kg;
* Imaging shows multiple cerebral infarction (low density > 1/3 brain hemisphere);
* The timing of stroke symptoms is not known;
* mRS score before stroke≥ 2 points;
* NIHSS score 1a (level of consciousness) ≥ 2 points during screening;
* CT/MRI imaging examination showed signs of intracranial hemorrhage or suspected subarachnoid hemorrhage despite CT/MRI imaging findings did not show abnormalities.
* Subjects have an acute bleeding tendency, including a platelet count of less than 100 × 109 / L, application of heparin or oral anticoagulant drugs (such as warfarin) within 24 hours before onset , and an INR > 1.6;
* Patients who are ready to go or have undergone endovascular treatment;
* Patients who had severe trauma or major surgery in the last 3 months (according to the investigator's assessment);
* A stroke has occurred in the last 3 months; or has a history of any stroke with diabetes;
* Severe liver damage, including liver failure, cirrhosis, portal hypertension (esophageal varices), and active hepatitis;
* Other diseases lead to patients with an expected survival time of no more than one year;
* Hypertension remains uncontrolled after active antihypertensive therapy. Uncontrolled hypertension refers to a systolic blood pressure >185 mmHg and/or a diastolic blood pressure >110 mmHg measured at intervals of at least 10mins, repeated 3 times;
* Blood glucose <50 mg/dl (equivalent to 2.78mmol/L) or >400 mg/dl (equivalent to 22.2mmol/L);
* Patients who are unable to cooperate or are unwilling to cooperate with epileptic seizures, or other mental illnesses during stroke episodes;
* Known to be allergic to research drugs or similar ingredients, or materials used in imaging studies;
* The restricted drug specified in the protocol or any drug that may interfere with the test results must be ingested or desired to continue to be ingested;
* Participating in other trials or has been participated in other trials within 30 days before randomization;
* Pregnancy or lactation, or women who have a positive pregnancy test result;
* The Subject who is unsuitable for this study in the opinion of the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-07-20 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with NIHSS score ≤1 or the decrease of 4 points or more from the baseline on the 14th day after treatment; | on the 14th day after treatment
  The National Institutes of Health Stroke Scale (NIHSS) is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items. The range of scores is from 0 (normal) to 42 (profound effect of stroke on patient).

SECONDARY OUTCOMES:
The proportion of subjects with NIHSS score ≤1 or the decrease of 4 points or more from the baseline at 72 hours after treatment; | at 72 hours after treatment;
  Proportion of patients with ≥4 point reduction in NIHSS or reaching 0-1 at 3 days (favourable clinical response) adjusted for baseline NIHSS and age.
The proportion of subjects with mRS score of 0-1 on the 30th day and 90th day after treatment; | on the 30th day and 90th day after treatment;
  The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0-5. A separate category of 6 is usually added for patients who expire. Standardized interviews to obtain a mRS score are recommended at 3 months (90 days) following hospital discharge.
  The scale runs from 0-5, running from perfect health without symptoms to Severe disability 0. -No symptoms.
  1. -No significant disability. Able to carry out all usual activities, despite some symptoms.
  2 .-Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. -Moderate disability. Requires some help, but able to walk unassisted.
  4. -Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. -Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
The proportion of subjects with mRS score of 0-2 on the 30th day and 90th day after treatment; | on the 30th day and 90th day after treatment;
Continuous changes of mRS scores on the 30th and 90th days after treatment; | on the 30th and 90th days after treatment;
The proportion of subjects with Barthel index score≥95 on the 30th day and 90th day after treatment; | on the 30th day and 90th day after treatment;
  The Barthel Index of Activities of Daily Living (ADLs) measures functional disability by quantifying patient performance in 10 activities of daily life. These activities can be grouped according to self-care (feeding, grooming, bathing, dressing, bowel and bladder care, and toilet use) and mobility (ambulation, transfers, and stair climbing). 5-point increments are used in scoring, with a maximal score of 100 indicating that a patient is fully independent in physical functioning, and a lowest score of 0 representing a totally dependent bed-ridden state.

OTHER OUTCOMES:
Percentage of subjects with symptomatic intracranial hemorrhage (sICH); | within 36h after thrombolysis
  sICH definition: 1、NINDS criteria: Any clinical deterioration within 36h after thrombolysis (NIHSS score point increase ≥ 1 point), imaging suggests intracranial hemorrhage; 2 、ECASS-II criteria: within 36h after thrombolysis, relative baseline or minimum NIHSS score point increase ≥ 4 points, The image suggests intracranial hemorrhage; 3、SITS criteria: within 36 hours after thrombolysis, the relative baseline or minimum NIHSS score point increased by ≥ 4 points, The image shows > 30% of the infarct area, there is a cerebral hematoma (PH-2 type). (This study will be evaluated and recorded according to the above three standards.
Mortality within 90 days after treatment; | within 90 days after treatment;
The Proportion of subjects with adverse events/serious adverse events within 90 days after treatment. | within 90 days after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li S, Wang X, Jin A, Liu G, Gu H, Li H, Campbell BCV, Fisher M, Yang Y, Wei Y, Wang J, Wang Y, Zhao X, Liu L, Li Z, Meng X, Wang Y. Safety and Efficacy of Reteplase Versus Alteplase for Acute Ischemic Stroke: A Phase 2 Randomized Controlled Trial. Stroke. 2024 Feb;55(2):366-375. doi: 10.1161/STROKEAHA.123.045193. Epub 2023 Dec 28. PMID 38152962